CLINICAL TRIAL: NCT07160036
Title: Exploring the Repeatability of Adaptive Optics Scanning Laser Ophthalmoscope Technology (AO-SLO Mona IIa) and the Differences in Cone Cell Density Between Individuals Who Undergone and Not Undergone Repeated Low-level Red-light
Brief Title: Repeatability of AO-SLO (Mona IIa) Technology and Cone Cell Density of Individuals Use Repeated Low-level Red-light Therapy
Acronym: AO-SLO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruihua Wei (Other)
Collaborators: Tianjin Medical University Eye Hospital (Other)
Responsible Party: Sponsor-Investigator, Ruihua Wei, Professor, Tianjin Medical University Eye Hospital
Organization: Tianjin Medical University Eye Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025YK-52
Record Dates: First submitted 2025-08-30; First posted 2025-09-08 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RLRL group (Experimental): Use RLRL (Model RS-200-2A, Eyerising; Suzhou Xuanjia Optoelectronic Technology Co., Ltd., Suzhou, China)
  Interventions: Device: RLRL(Model RS-200-2A, Eyerising; Suzhou Xuanjia Optoelectronic Technology Co., Ltd., Suzhou, China))
- No RLRL Group (No Intervention): No use RLRL

INTERVENTIONS:
Device: RLRL(Model RS-200-2A, Eyerising; Suzhou Xuanjia Optoelectronic Technology Co., Ltd., Suzhou, China)) — use RLRL twice a day
  Arms: RLRL group

SUMMARY:
To explore the repeatability of AO-SLO (Mona IIa) technology and the difference of cone cell density between individuals who used or not used repeated low-intensity red light treatment

DETAILED DESCRIPTION:
This study focuses on the population with long-term use of repetitive low-intensity myopia, exploring the safety of repetitive low-intensity red light over a long period of use, and providing data support and clinical guidance for the field of repetitive low-intensity red light. It investigates the repeatability of adaptive optics scanning laser ophthalmoscope technology and observes the safety of repetitive low-intensity red light treatment for children over a long period of use.

ELIGIBILITY:
Inclusion Criteria:

* 6 - 55 years old, gender not limited; Obtained informed consent.

Exclusion Criteria:

* Children with obvious strabismus and amblyopia
* With congenital eye disease, such as congenital cataract, congenital retinal disease
* Secondary myopia (such as premature retinopathy or other eye diseases in infants and children caused secondary myopia), or myopia combined with systemic syndrome (such as Marfan syndrome)
* Had internal eye surgery (such as cataract extraction, intraocular lens implantation, anti-glaucoma surgery, etc.)
* Refractive medium opacity (such as corneal disease, crystal opacity, etc.)
* Bnormal intraocular pressure and clinical significance (IOP <10 mmHg or IOP>21mmHg or binocular IOP difference ≥5mmHg)
* Fundus chorioretinopathy (except for high myopia fundus degenerative changes) or other intraocular diseases
* Optic nerve damage or congenital optic nerve dysfunction
* Can not be regularly checked
* The adjustment range is less than 8D or obvious near difficulties
* Other reasons researchers think it is not suitable for inclusion in researchers

Ages: 6 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
The density of cone cells | From enrollment to the end of treatment at 3 weeks

SECONDARY OUTCOMES:
Repeatability of adaptive optics scanning laser ophthalmoscope technology of cone cell density | From enrollment to the end of treatment at 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Wei, Principal Investigator — Tianjin Medical University Eye Hospital, Tianjin, Tianjin 120120 Recruiting
Locations (1):
- Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No